CLINICAL TRIAL: NCT05011838
Title: A Multi-component Intervention to Reduce Gaps in Hypertension Care and Control in Medellin, Colombia
Brief Title: Evaluation of the Effectiveness of an Intervention to Reduce Gaps in Hypertension Care in Low-income Medellin, Colombia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the devasting impact of Covid-19 on Colombian health services, the execution of the study was halted shortly after all involved actors had been trained
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University Ghent (Other); Facultad Nacional de Salud Publica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1294/19
Record Dates: First submitted 2021-08-06; First posted 2021-08-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
Keywords: Heart Disease Risk Factors; Primary Health Care; Controlled Before-After Studies; Latin America; Colombia
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Two deprived Communes of the city have been selected as intervention and control arms. All the intervention components will be implemented in Commune 2, located in the northeast of Medellin. Commune 6, located northwest of Medellin, has been selected as the control area to deliver routine care. Two representative population surveys of adults aged 35 years or older will be undertaken in the intervention and the control Communes two years apart, one before the intervention implementation and the other after. The surveys will randomly include different individuals. The main outcomes assessed will be the gaps in hypertension diagnosis, treatment, follow-up and control.
Who Masked: Participant
Masking Description: Participants are kept unaware of the intervention implementation and its assignment in one commune or another. Furthermore, participants will be randomly recruited in both communes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A multi-component intervention to improve hypertension care and control (Experimental): The intervention will be implemented in Commune 2. It will integrate activities related to 1) Health services redesign, 2) Clinical staff training and 3) Patient and community engagement. The intervention activities will be implemented by health services staff with technical assistance from the investigation team.
  Interventions: Other: 1. Health Services Redesign; Other: 2. Clinical Staff Training; Other: 3. Patient and Community Engagement
- Routine Care (No Intervention): The Commune 6 was selected as control area, where routine care will be delivered.

INTERVENTIONS:
Other: 1. Health Services Redesign — 1.1. Healthy Hearts service: a nursing station providing blood pressure measurement, cardiovascular risk assessment, preventive counselling and effective follow-up in extended opening hours.
  1.2. Hypertension screening: All adults attending health care facilities who did not have their blood pressure measured in the previous year will be referred to the Healthy Hearts Service for screening.
  1.3. Clinical management: 1.3.1. Creation of the cardiovascular risk team: a group of doctors supervising hypertension management and coordinating improvement.
  1.3.2. Guideline-based standardized diagnostic and treatment protocols: a simplified diagnostic and treatment algorithm will identify a core set of primary and secondary antihypertensive medications.
  1.3.3. Availability of antihypertensive medications: it will be assured through procurement mechanisms and its availability will be communicated to clinicians at the beginning of each week and ad hoc in case of stock-outs.
  Arms: A multi-component intervention to improve hypertension care and control
Other: 2. Clinical Staff Training — 2.1. Training on good clinical management of hypertension: focused on correct blood pressure measurement, use of evidence-based guidelines, cardiovascular risk assessment, use of a standardized diagnostic and treatment algorithm, correct prescription of pharmacological and non-pharmacological treatment, patient counselling, and how to tackle clinical inertia.
  2.2. Training on communication skills and patients' needs assessment for all health workers involved in hypertension care. This training will be designed under the "patient-centred medicine" framework, aiming at equipping health providers with tools for understanding patients' feelings and experience of illness, and to improve their capacity to address social, psychological, and behavioural dimensions of hypertension care.
  Arms: A multi-component intervention to improve hypertension care and control
Other: 3. Patient and Community Engagement — 3.1. Patient empowerment: "expert hypertensive patients" , under the supervision of a social worker, will provide support and transmit their know-how to other patients in need, particularly those newly diagnosed or non-adherent to treatment or presenting uncontrolled hypertension.
  3.2. Community engagement: a Community Hypertension Outreach Group will be set up, composed of existing voluntary community health workers, who will be trained and certified. This group will conduct blood pressure measurements in selected public areas of the commune, referring those with positive screening to the nearest health facility for diagnosis confirmation. It will also provide health information with emphasis on healthy lifestyles. Existing local communication channels such as the community radio and the local newspaper will be engaged.
  Arms: A multi-component intervention to improve hypertension care and control

SUMMARY:
This study evaluates the effectiveness of a multi-component intervention to reduce the gaps in hypertension care and control at a population level in low-income Communes of Medellin, Colombia, and assess the process and fidelity of the intervention's implementation.

DETAILED DESCRIPTION:
A multi-component intervention was designed based on international guidelines, a cross-sectional population survey results, and consultation with the community and institutional stakeholders. Three main components integrate activities related to (I) Health services redesign, (II) Clinical staff training (III) Patient and community engagement. The effectiveness of the intervention will be evaluated in a controlled before-after quasi-experimental study, with two deprived Communes of the city selected as intervention and control arms. Two representative population-based surveys of adults aged 35 years or older will be undertaken in the intervention and the control Communes two years apart, one before the intervention implementation and the other after. The surveys will include different adults. The main outcomes assessed will be the gaps in hypertension diagnosis, treatment, follow-up and control. Effectiveness will be evaluated with "difference in difference" measures. Generalized estimation equations models will be fitted considering the clustered nature of data and adjusting for potential confounding variables. The implementation process will be studied with mixed methods. Finally, implementation fidelity will be documented to assess to which degree the components of the intervention were implemented as intended.

ELIGIBILITY:
Inclusion Criteria:

* 35 years or older
* Permanent inhabitant of the selected Communes
* Must be able to provide written informed consent

Exclusion Criteria:

* Mental disability
* Unable to answer the questionnaire

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-14 (Estimated); Primary Completion 2025-02-14 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Number of individuals self-reporting a previous diagnosis of hypertension and encountered with uncontrolled hypertension during the study. | through the population survey completion, up to 2 months
  Uncontrolled hypertension: an average blood pressure measurement higher than 140/90 mmHg for aware hypertensive patients between 35 and 59 years old or for diabetic patients regardless of age, and higher than 150/90 mmHg for aware hypertensive patients aged 60 years or older.

SECONDARY OUTCOMES:
Number of individuals without a previous diagnosis but presenting hypertension during the study. | through the population survey completion, up to 2 months
  Hypertension: an average repeat blood pressure measurement equal to or higher than 140/90 mmHg.
Number of individuals self-reporting a previous diagnosis of hypertension who did not attend a follow-up consultation during the last year. | through the population survey completion, up to 2 months
  Aware hypertensive individuals who self-report that they did not attend a follow-up consultation for hypertension during the last year.
Number of aware hypertensive individuals who received a prescription of antihypertensive medication but either do not take the drugs or are non-adherent. | through the population survey completion, up to 2 months
  Patients with a prescription of antihypertensive medication who self-report that they do not take the drugs or, assessed by mean of the 4-item Medication Adherence Questionnaire, are non-adherent.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban A Londoño-Agudelo, MD.MPH., Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium; Patrick Van der Stuyft, MD.MPH.PhD, Study Director — University Ghent
Locations (1):
- Unidad Hospitalaria de Santa Cruz, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data sets, properly anonymized, underlying our publications of research results, will be shared upon reasonable and formal institutional request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The investigators plan to publish the research protocol, which would be available in November 2021. Participant data sets underlying our results would be available starting 2 months after publication.
Access Criteria: The study protocol and the corresponding statistical analysis plan will be broadly available after its publication planned for November 2021. Other supporting information will be shared only with accredited scientific researchers through an institutional formal request via email and confirmed by phone. Requests for data sharing must comply legal regulations in Colombia and have the endorsement of the Institutional Research Board of the Antwerp Institute of Tropical Medicine.

REFERENCES:
- [Background] Londono Agudelo E, Garcia Farinas A, Perez Ospina V, Taborda Perez C, Villacres Landeta T, Battaglioli T, Gomez Arias R, Van der Stuyft P. Out-of-pocket expenditure for hypertension care: a population-based study in low-income urban Medellin, Colombia. Glob Health Action. 2020 Dec 31;13(1):1806527. doi: 10.1080/16549716.2020.1806527. PMID 32867605
- [Background] Londono Agudelo E, Perez Ospina V, Battaglioli T, Taborda Perez C, Gomez-Arias R, Van der Stuyft P. Gaps in hypertension care and control: a population-based study in low-income urban Medellin, Colombia. Trop Med Int Health. 2021 Aug;26(8):895-907. doi: 10.1111/tmi.13599. Epub 2021 May 22. PMID 33938098
- [Derived] Londono Agudelo EA, Battaglioli T, Soto A, Vasquez Gomez J, Aguilar Ramirez H, Perez Ospina V, Rodriguez Salva A, Ortiz Solorzano P, Perez D, Gomez-Arias R, Van Der Stuyft P. Protocol for a controlled before-after quasi-experimental study to evaluate the effectiveness of a multi-component intervention to reduce gaps in hypertension care and control in low-income communes of Medellin, Colombia. BMJ Open. 2022 Aug 24;12(8):e056262. doi: 10.1136/bmjopen-2021-056262. PMID 36002215

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT05011838/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT05011838/ICF_001.pdf